CLINICAL TRIAL: NCT00583037
Title: FEASIBILITY OF 24 Hrs VENTILATION WITH NEURALLY ADJUSTED VENTILATORY ASSIST (NAVA) IN PATIENTS WITH ACUTE RESPIRATORY FAILURE
Brief Title: 24-Hour NAVA Ventilation in Acute Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Fabrice Brunet, St. Michael's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 05-242
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2009-06-01 (Estimated); Status verified 2009-05

CONDITIONS: Respiration, Artificial; Respiratory Insufficiency
Keywords: Neurally Adjusted Ventilatory Assist; Sleep quality; Adult; Critical Care
MeSH Terms: conditions — Respiratory Aspiration; Respiratory Insufficiency; Sleep Initiation and Maintenance Disorders | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NAVA (Experimental): Implementation of NAVA for 24 hours
  Interventions: Device: Neurally Adjusted Ventilatory Assist (NAVA)

INTERVENTIONS:
Device: Neurally Adjusted Ventilatory Assist (NAVA) — Mechanical ventilation controlled by diaphragm electrical activity
  Other Names: Servo i Ventilator System- NAVA Catheters (6671277, 6671280, 6671282, 6671287, 6671290); Servo i Ventilator System- NAVA HW option (6671957); Servo i Ventilator System- NAVA SW option (6671965)

SUMMARY:
Neurally Adjusted Ventilatory Assist (NAVA) is a new mode of mechanical ventilation that is controlled by the electrical activity of the diaphragm (EAdi). The EAdi is a signal that represents the patient's breathing effort, and hence with NAVA, the assist being delivered is synchronized and proportional to the demands of the patient. This is a prospective physiological study of the feasibility of NAVA ventilation over 24 hours. The aim is to demonstrate that NAVA can maintain spontaneous breathing and unload the respiratory muscles during both sleep and wake cycles over a 24 hour period.

DETAILED DESCRIPTION:
To date, studies using NAVA technology have been limited to short term evaluations (under 3 hours). No serious adverse events have been observed in patients enrolled in our 3-hour study of NAVA in patients with acute lung injury. All 15 patients successfully tolerated the period of ventilation (i.e. there were no dropouts) with NAVA and the stability of the blood gas parameters over time reveals the efficiency of this new mode of ventilation in regards to oxygenation.

A longer study may help to evaluate patient tolerance of NAVA and stability over time. A longer study will also demonstrate the feasibility of NAVA to adapt to changes in respiratory drive, changes in patient status, and the interventions of health care providers. A longer time frame should help us understand the parameters for titration of NAVA settings over time and establish some indications/limits for the future use of this promising technique. This intermediate study will generate the data necessary for the development of additional protocols to refine NAVA application and to compare NAVA to other assist modes.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU will be screened on a daily basis for the presence of the following characteristics:
* Adult (>18 years old) intubated and mechanically ventilated patients with evidence of spontaneous breathing defined as:

  1. Patient is on pressure support ventilation OR
  2. Patient is on pressure control ventilation with the ability to trigger 50% of the breaths.
* Sedation Agitation Score (SAS) score greater than or equal to 2
* Presence of an arterial line
* Patients meeting these criteria will be considered eligible for recruitment into the study

General Exclusion Criteria:

* Next of kin unavailable
* Patient/next of kin refuses informed consent.
* Attending physician refuses to allow enrollment
* Pregnancy

Exclusion Criteria Related to the Technique:

* Any contraindication to insertion of a nasogastric tube including, but not limited to: severe oropharyngeal malformation or bleeding, esophageal varices, tumor, infection, stenosis, or rupture
* Hemophilia or other severe bleeding disorder
* Presence or suspicion of central/brain stem neurologic disorder/severe neuromuscular disease
* Treatment with neuromuscular blockers
* History of heart and/or lung transplantation

Exclusion Criteria Related to the Clinical Stability of the Patient:

* Mean arterial blood pressure < 60 mm Hg with or without vasopressors or inotropes
* Any contraindication to reducing sedation to obtain a targeted SAS score of 3 (e.g. anticipated hemodynamic instability after reduction of sedation)
* Patients with evidence of any of the above exclusions will not be eligible for enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-05; Primary Completion 2008-01 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of NAVA as assessed by: • Assessment of FiO2 changes • Assessment of the NAVA catheter function: o Stability of the EAdi signal from NAVA catheter o Requirements for NAVA catheter position change • Reasons for ventilator alarms | 24 hours

SECONDARY OUTCOMES:
Patient tolerance of NAVA as assessed by: • Changes in SAS scoring and sedation requirement • Changes in vital signs (HR/BP) and vasopressors requirements • Changes in oxygenation/ventilation | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Brunet, MD, Principal Investigator — Unity Health Toronto; Christer Sinderby, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St-Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Sinderby C, Navalesi P, Beck J, Skrobik Y, Comtois N, Friberg S, Gottfried SB, Lindstrom L. Neural control of mechanical ventilation in respiratory failure. Nat Med. 1999 Dec;5(12):1433-6. doi: 10.1038/71012. No abstract available. PMID 10581089
- [Background] Sinderby C. Ventilatory assist driven by patient demand. Am J Respir Crit Care Med. 2003 Oct 1;168(7):729-30. doi: 10.1164/rccm.2307004. No abstract available. PMID 14522808
- [Background] Beck J, Brander L, Slutsky AS, Reilly MC, Dunn MS, Sinderby C. Non-invasive neurally adjusted ventilatory assist in rabbits with acute lung injury. Intensive Care Med. 2008 Feb;34(2):316-23. doi: 10.1007/s00134-007-0882-x. Epub 2007 Oct 25. PMID 17960364
- [Background] Beck J, Campoccia F, Allo JC, Brander L, Brunet F, Slutsky AS, Sinderby C. Improved synchrony and respiratory unloading by neurally adjusted ventilatory assist (NAVA) in lung-injured rabbits. Pediatr Res. 2007 Mar;61(3):289-94. doi: 10.1203/01.pdr.0000257324.22406.93. PMID 17314685
- [Background] Allo JC, Beck JC, Brander L, Brunet F, Slutsky AS, Sinderby CA. Influence of neurally adjusted ventilatory assist and positive end-expiratory pressure on breathing pattern in rabbits with acute lung injury. Crit Care Med. 2006 Dec;34(12):2997-3004. doi: 10.1097/01.CCM.0000242520.50665.9F. PMID 16957635